CLINICAL TRIAL: NCT03933943
Title: A Phase 1, Randomized, Placebo-Controlled, Multiple- Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous LY3361237 in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of LY3361237 in Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17180; I9S-MC-BTAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-04-30; First posted 2019-05-01 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03-01

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3361237 (Experimental): LY3361237 administered subcutaneously (SC)
  Interventions: Drug: LY3361237
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3361237 — Administered SC
  Arms: LY3361237
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety of LY3361237 and any side effects that might be associated with it when given to participants with systemic lupus erythematosis (SLE). LY3361237 will be administered by injections just under the skin. The study will last up to 26 weeks and may include up to 17 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have received a diagnosis of SLE at least 24 weeks before screening (at least 4 of 11 criteria in 1997 revised American College of Rheumatology [ACR] classification)
* If a participant is taking oral prednisone (or prednisone equivalent) for SLE, the dose must be ≤20 milligrams per day (mg/day) for at least 8 weeks prior to screening, and must have been stable for at least the last 2 weeks
* If a participant is taking any of the following medications for SLE, the medication must have been used for at least 12 weeks and stable for at least the last 8 weeks:

  * Azathioprine ≤200 mg/day
  * Antimalarial (e.g., chloroquine, hydroxychloroquine, quinacrine)
  * Mycophenolate mofetil ≤2 g/day or mycophenolic acid ≤1.44 grams per day (g/day)
  * Oral, SC, or intramuscular methotrexate ≤15 milligrams per week (mg/week)

Exclusion Criteria:

* Participants must not have a history of, or current, inflammatory joint or skin disease other than SLE
* Participants must not have a current active bacterial, viral, or fungal infection
* Participants must not have evidence of significant liver or kidney dysfunction
* Participants must not have received cytotoxic medications (e.g., cyclophosphamide) within the last 3 months.
* Participants must not have received any intra-articular, intramuscular, or intravenous glucocorticoids within the last 3 months
* Participants must not have received blood products (e.g., blood transfusion, platelets, etc.) within the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline through Day 155
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3361237 | Day 1 predose through Day 155
  PK: Cmax of LY3361237
PK: Area Under the Concentration Versus Time Curve (AUC) Over the Dosing Interval of LY3361237 | Day 1 predose through Day 155
  PK: AUC Over the Dosing Interval of LY3361237

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - Pinnacle Research Group, Anniston, Alabama
  - Clinical Research of West Florida, Clearwater, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - North Georgia Rheumatology, PC, Lawrenceville, Georgia
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Accurate Clinical Management LLC - Katy, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3361237 in Participants With Systemic Lupus Erythematosus — https://trials.lillytrialguide.com/en-US/trial/eiRWT5wAOkRpZOHEo4Ira